CLINICAL TRIAL: NCT03010878
Title: Yoga and Occupational Therapy to Improve Pain
Acronym: YoPain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Responsible Party: Principal Investigator, Arlene Schmid, Associate Professor, Colorado State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15.6017H
Record Dates: First submitted 2016-12-29; First posted 2017-01-05 (Estimated); Results first posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Chronic Pain
Keywords: yoga; chronic pain; occupational therapy; self-management
MeSH Terms: conditions — Chronic Pain | interventions — Yoga; Self-Management

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Yoga Arm (Experimental): Yoga administered twice a week for 8 weeks. Self-management education sessions administered once a month through the University of Colorado Health Fort Collins Family Medicine Residency Program Pain Management Clinic (Pain Clinic). Yoga interventions were administered twice a week at the Pain Clinic.
  Interventions: Other: Yoga; Other: Self-management
- Wait-list Control Arm (Experimental): Participants received only self-management intervention, which is provided once a month through the University of Colorado Health Fort Collins Family Medicine Residency Program Pain Management Clinic.
  Interventions: Other: Self-management

INTERVENTIONS:
Other: Yoga — The yoga intervention group addressed pain as a primary variable and balance as a secondary variable and how to best manage these symptoms in the clinic and community.
  Yoga was delivered in sitting, standing, and floor postures
  Arms: Yoga Arm
Other: Self-management — The self-management education group was provide once a month through University of Colorado Health Fort Collins Family Medicine Residency Program Pain Management Clinic. The program consisted of lifestyle variations, accountability, modifications, and strategies to management pain in daily life.

SUMMARY:
This was a randomized control trial of a yoga and self-management intervention for individuals with chronic pain. Participants were assigned to either a wait-list control group (self-management only), or a yoga intervention (self-management and yoga). Self-management education session occurred monthly within the community. Group yoga intervention was delivered two times a week with a specifically designed program that was progressively more difficult. Assessments were then administered pre and post intervention, and a semi-structured interview was completed following the intervention. Quantitative and qualitative data were then compared between groups.

DETAILED DESCRIPTION:
This was a randomized control trial completed with two specific aims.

Aim 1: To assess the feasibility of completing a group yoga intervention in conjunction with an ongoing self-management education for people with chronic pain.

Aim 2: To explore the preliminary efficacy of a group yoga intervention in people with chronic pain. The key variables of interest were pain interference, functional performance, balance, strength, mobility, and quality of life (QoL)

ELIGIBILITY:
Inclusion Criteria:

* greater than 18 years of age
* Individual with self-reported pain for over six months
* attending outpatient pain clinic
* ability to attend yoga classes
* ability to complete assessments
* ability to provide informed consent

Exclusion Criteria:

* consistent yoga practice over the past year
* self-reported exercise restrictions
* serious and recent medical procedures or conditions without doctor's note
* high risk pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2015-08; Primary Completion 2016-05 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arlene Schmid, PhD, Principal Investigator — Colorado State University
Locations (1):
- UC Health Fort Collins Family Medicine Residency Program Pain Management Clinic, Fort Collins, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schmid AA, Atler KE, Malcolm MP, Grimm LA, Klinedinst TC, Marchant DR, Marchant TP, Portz JD. Yoga improves quality of life and fall risk-factors in a sample of people with chronic pain and Type 2 Diabetes. Complement Ther Clin Pract. 2018 May;31:369-373. doi: 10.1016/j.ctcp.2018.01.003. Epub 2018 Feb 15. PMID 29526474

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment completed - all completed at a pain clinic
Groups:
- Yoga Arm: Yoga administered twice a week for 8 weeks. Self-management education sessions administered once a month through the University of Colorado Health Fort Collins Family Medicine Residency Program Pain Management Clinic (Pain Clinic). Yoga interventions were administered twice a week at the Pain Clinic.
  Yoga: The yoga intervention group addressed pain as a primary variable and balance as a secondary variable and how to best manage these symptoms in the clinic and community.
  Yoga was delivered in sitting, standing, and floor postures
  Self-management: The self-management education group was provide once a month through University of Colorado Health Fort Collins Family Medicine Residency Program Pain Management Clinic. The program consisted of lifestyle variations, accountability, modifications, and strategies to management pain in daily life.
Period: Overall Study
Arm/Group | Yoga Arm | Wait-list Control Arm
Started | 44 | 39
Completed | 28 | 39
Not Completed | 16 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Yoga Arm | Wait-list Control Arm | Total
Number analyzed (Participants) | 28 | 39 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.04 (9.6) | 49.15 (10.82) | 50.78 (10.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 27 | 46
  Male | 9 | 12 | 21
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 28 | 39 | 67
Brief Pain Inventory [Mean (Standard Deviation); unit: units on a scale] — Scale is measured from 0-10, with a higher score indicating worse pain severity and interference on everyday life.
  units on a scale | 7.05 (1.22) | 6.39 (1.53) | 6.72 (1.37)

OUTCOME MEASURES:

1. Primary Outcome: Brief Pain Inventory--Short Form
Description: The Brief Pain Inventory (Short Form) is a 9 item self-report questionnaire designed to assess general pain. Minimum 0 - Maximum 10 (higher score is indicated worse severity and interference with everyday life).
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Yoga Arm | Wait-list Control Arm
Number analyzed (Participants) | 28 | 39
units on a scale | 7.05 (1.22) | 6.39 (1.53)

ADVERSE EVENTS:
Time Frame: Participants were monitored for adverse events for the full duration of the study - 1 year.
Description: Both groups had adverse events monitored throughout the study. The waitlist cohort was offered yoga for up to 16 weeks, however, the primary endpoint was measured after 8 weeks of yoga/waitlist control. All adverse events are reflected in the chart below.
Arm/Group | Yoga Arm | Wait-list Control Arm
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/39
Other Adverse Events (participants affected / at risk) | 0/28 | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes